CLINICAL TRIAL: NCT01540370
Title: Study Comparing Quantitative Assessments in Open-angle Glaucoma (OAG) and/or Ocular Hypertension (OHT)
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: 192024-076
Record Dates: First submitted 2012-02-23; First posted 2012-02-28 (Estimated); Results first posted 2013-09-19 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-07

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with OAG and/or OHT: Patients with OAG and/or OHT
  Interventions: Other: No Treatment

INTERVENTIONS:
Other: No Treatment — No treatment

SUMMARY:
This study will evaluate assessments from the Goniometric Lens compared with those from anterior segment imaging in patients with open-angle glaucoma (OAG) and/or ocular hypertension (OHT).

ELIGIBILITY:
Inclusion Criteria:

* Open-angle glaucoma or ocular hypertension

Exclusion Criteria:

* Allergy or sensitivity to diagnostic agents used in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with open-angle glaucoma and/or ocular hypertension
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2012-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients With OAG and/or OHT
Started | 102
Completed | 100
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Patients With OAG and/or OHT
Number analyzed (Participants) | 102
Age Continuous [Mean (Standard Deviation); unit: Years] | 64.1 (12.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 49

OUTCOME MEASURES:

1. Primary Outcome: Intra- Examiner Agreement in Angle Width by Goniometric Lens
Description: Intra-rater agreement (for each of the 6 raters) of Large Step angle width (range: 0.5 to 5.5 with 0.5 unit intervals) was evaluated using weighted kappa (Fleiss-Cohen) statistics. The angle is the area between the iris and cornea of the eye. Each examiner performed a pair of angle-width measurements by goniometric lens predilation (ie, 2 measurements per examiner). The degree of agreement within raters was interpreted according to Landis and Koch, where: <0:poor, 0.00-0.20:slight, 0.21-0.40:fair, 0.41-0.60:moderate, 0.61-0.80:substantial, and 0.81-1.00:almost perfect.
Time Frame: Day 1
Population: Modified Intent to Treat: enrolled patients with unobstructed and measurable inferior angles by goniometric reading and anterior segment optical coherence tomography (OCT)
Measure: Number; unit: Kappa statistics
Arm/Group | Patients With OAG and/or OHT
Number analyzed (Participants) | 100
Kappa statistics | 0.88

2. Primary Outcome: Inter- Examiner Agreement in Angle Width by Goniometric Lens
Description: Inter-rater agreement (among 6 raters) of Large Step angle width (range: 0.5 to 5.5 with 0.5 unit intervals) was evaluated using weighted kappa (Fleiss-Cohen) statistics. The angle is the area between the iris and cornea of the eye. Each examiner performed a pair of angle-width measurements by goniometric lens predilation (ie, 2 measurements per examiner). The degree of agreement within raters was interpreted according to Landis and Koch, where: <0:poor, 0.00-0.20:slight, 0.21-0.40:fair, 0.41-0.60:moderate, 0.61-0.80:substantial, and 0.81-1.00:almost perfect.
Time Frame: Day 1
Population: as for outcome 1
Measure: Number; unit: Kappa statistics
Arm/Group | Patients With OAG and/or OHT
Number analyzed (Participants) | 100
Kappa statistics | 0.72 [0.51 to 0.85]

ADVERSE EVENTS:
Description: The Safety Population is used to assess all Serious Adverse Events (SAEs) and Adverse Events (AEs). The Safety Population includes all enrolled patients who have been examined in the study eye.
Arm/Group | Patients With OAG and/or OHT
Serious Adverse Events (participants affected / at risk) | 0/101
Other Adverse Events (participants affected / at risk) | 0/101

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.